CLINICAL TRIAL: NCT02921568
Title: Side-by-Side Comparison of P200TE and Spectral OCT/SLO on Diseased Eyes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Optos, PLC (Industry)
Collaborators: Optos, Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: OPT1018
Record Dates: First submitted 2016-09-16; First posted 2016-10-03 (Estimated); Last update posted 2017-03-14 (Actual); Status verified 2016-09

CONDITIONS: Retinal Disease; Glaucoma
MeSH Terms: conditions — Retinal Diseases; Glaucoma

ARMS (1):
- All patients (Other): All patients will be imaged on the P200TE and Spectral OCT/SLO devices.
  Interventions: Device: P200TE; Device: Spectral OCT/SLO

INTERVENTIONS:
Device: P200TE — Optical Coherence Tomography and Scanning Laser Ophthalmoscope device.
Device: Spectral OCT/SLO — Optical Coherence Tomography and Scanning Laser Ophthalmoscope device.

SUMMARY:
This study is designed to evaluate and compare in-tissue performance of OCT scans on the new Optos P200TE, versus the predicate Optos Spectral OCT/SLO device.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects 18 years of age or older who have full legal capacity to volunteer;
2. Subjects who have signed the informed consent;
3. Subjects who can follow the instructions by the clinical staff at the clinical site, and can attend examinations on the scheduled examination date;
4. Subjects who agree to participate in the study;
5. Subjects with current BSCVA 20/400 or better in the ocular disease study eye(s);
6. Subjects diagnosed with ocular disease including but not limited to: Macular Degeneration, Diabetic Macular Edema, Diabetic Retinopathy, Central Serous Retinopathy, Macular Hole, Epiretinal Membrane, Macular Edema, Glaucoma, and others in the retinal disease study eye(s) as confirmed at the study visit or within the past six (6) months.

Exclusion Criteria:

1. Subjects unable to tolerate ophthalmic imaging;
2. Subjects with ocular media not sufficiently clear to obtain acceptable OCT images;
3. Subjects without ocular disease in study eye(s), as determined by self-report and/or investigator assessment at the study visit;
4. Subjects with history of leukemia, dementia or multiple sclerosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-09; Primary Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
retinal thickness | completion of the study, up to 5 years
Retinal Nerve Fibre Layer Thickness | completion of the study, up to 5 years
Optic Nerve Head Topography | completion of the study, up to 5 years
Cup/Disc Ratio | completion of the study, up to 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Center Ophthalmology Associates, San Antonio, Texas, United States